CLINICAL TRIAL: NCT05217940
Title: The Effectiveness of Screening Women With Lower Genital Tract Neoplasia or Cancers for Anal Cancer Precursors
Brief Title: Screening Women With Prior HPV for Anal Neoplasia
Acronym: SWAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Keith M Sigel, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GCO 20-0309
Record Dates: First submitted 2022-01-14; First posted 2022-02-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HPV-related Lower Genital Tract Neoplasias; HPV-related Anal Neoplasias; Early Stage Lower Genital Tract Cancers
Keywords: anal cancer; anal precancerous; anal high grade intraepithelial lesion; anal cytology; high resolution anoscopy; anal human papilloma virus testing
MeSH Terms: conditions — Anus Neoplasms | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Women With Prior HPV for Anal Neoplasia (Experimental): Standard of care anal cancer screening with anal cytology, HPV testing and high resolution anoscopy.
  Interventions: Diagnostic Test: Diagnostic tests for anal cancer screening

INTERVENTIONS:
Diagnostic Test: Diagnostic tests for anal cancer screening — The initial screening interventions will include the collection of (1) anal cytology; (2) self-collected HPV testing specimens (by subjects); (3) a clinician collected HPV specimen. A digital rectal exam will also be done on all patients.

SUMMARY:
The goal of this single arm trial is to prospectively evaluate screening methods for anal cancer precursors in HIV uninfected women with a history of lower genital tract neoplasias and cancers.

DETAILED DESCRIPTION:
This single arm trial will enroll 300 HIV uninfected women with a history of genital neoplasia (ie., cervical intraepithelial neoplasia grade 2-3, vaginal intraepithelial neoplasia grade 2-3 or vulvar intraepithelial neoplasia grade 2-3) or early stage cervical or vulvar cancer to evaluate the test characteristics of anal cancer screening tests (cytology, HPV testing and high resolution anoscopy) and determine the prevalence and incidence of anal high-grade squamous intraepithelial lesions in this population. Participants will undergo evaluation at baseline and then at 12 and 24 months. The investigators will also measure the acceptability of anal cancer screening in this previously unstudied group. The trial is expected to run from 2021-2027.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of pathologically proven high-grade genital HPV-associated neoplastic disease (cervical intraepithelial neoplasia 2+, vulvar intraepithelial neoplasia 2+, or vaginal intraepithelial neoplasia 2+, or history of non-metastatic cervical, vaginal or vulvar cancer)
* Documented HIV seronegativity
* Aged 35 years and older
* Seen in the Mount Sinai Health System (MSHS) or the Harris Health System (HHS) in Houston
* English or Spanish speaking

Exclusion Criteria:

• prior history or high resolution anoscopy

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of anal cytology | Baseline
  Test sensitivity and specificity

SECONDARY OUTCOMES:
Concordance of self- and clinician-collected PCR testing | baseline
  Proportionate concordance of high-risk HPV testing
Prevalence of hrHPV types at baseline | Baseline
  Proportion of subjects with high-risk HPV and subtype proportions
hrHPV with Cobas PCR testing (self-collected) | Baseline
  Presence of high-risk HPV subtype
hrHPV with Cobas PCR testing (self-collected) | 12 months
  Presence of high-risk HPV subtype
hrHPV with Cobas PCR testing (self-collected) | 24 months
  Presence of high-risk HPV subtype
hrHPV with Cobas PCR testing (clinician-collected) | Baseline
  Presence of high-risk HPV subtype
hrHPV with Cobas PCR testing (clinician-collected) | 12 months
  Presence of high-risk HPV subtype
hrHPV with Cobas PCR testing (clinician-collected) | 24 months
  Presence of high-risk HPV subtype
Prevalence of aHSIL at baseline | Baseline
  Proportion of subjects with aHSIL
Incidence of aHSIL at follow-up | 24 months
  Proportion of subjects with new aHSIL during follow-up period
Screening Experience Survey | Baseline
  Survey measures anal cancer screening test acceptability. Each item is scored 0-3, with higher score indicting more acceptability. 0-3. There is no total scale. Each question is scored separately and the overall results are used qualitatively.
Incidence of hrHPV, by type | 12 months
  Proportion of subjects with new hrHPV infection
Incidence of hrHPV, by type | 24 months
  Proportion of subjects with new hrHPV infection
Proportion of subjects with new hrHPV infection | 12 months
  Proportion of subjects with prevalent hrHPV without measurable hrHPV at follow-up
Proportion of subjects with new hrHPV infection | 24 months
  Proportion of subjects with prevalent hrHPV without measurable hrHPV at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sigel, MD, PhD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Elizabeth Chiao, MD, Principal Investigator — M.D. Anderson Cancer Center; Ashish Deshmukh, PhD, Principal Investigator — Medical University of South Carolina
Locations (3):
- United States (3):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Email principal investigator: keith.sigel@mssm.edu